CLINICAL TRIAL: NCT05270408
Title: Noninvasive Brain Stimulation in Mild Cognitive Impairment and Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Christian Lobue, ASSISTANT PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU-2021-0974
Record Dates: First submitted 2021-12-30; First posted 2022-03-08 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia
Keywords: Transcranial direct current stimulation; Alzheimer Disease; Mild Cognitive Impairment; Dementia; MCI; Mild neurocognitive disorder; Amnestic; Pre- alzheimer
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Active stimulation at 1mA (Experimental): Participants will receive 1 mA active HD-tDCS for 20 minutes.
  Interventions: Device: Active Transcranial direct current stimulation (STARStim 8)
- Active stimulation at 2mA (Experimental): Participants will receive 2 mA active HD-tDCS for 20 minutes.
  Interventions: Device: Active Transcranial direct current stimulation (STARStim 8)
- Sham group (Sham Comparator): Participants will receive sham HD-tDCS for 20 minutes, meaning no stimulation.
  Interventions: Device: Sham Transcranial direct current stimulation (STARStim 8)

INTERVENTIONS:
Device: Active Transcranial direct current stimulation (STARStim 8) — Participants wear a neoprene cap on their head and electrodes filled with gel are attached and will deliver 1mA to the scalp.
  Arms: Active stimulation at 1mA
Device: Active Transcranial direct current stimulation (STARStim 8) — Participants wear a neoprene cap on their head and electrodes filled with gel are attached and will deliver 2mA to the scalp.
  Arms: Active stimulation at 2mA
Device: Sham Transcranial direct current stimulation (STARStim 8) — Participants wear a neoprene cap on their head and electrodes filled with gel are attached and will deliver no current to the scalp.
  Arms: Sham group

SUMMARY:
The research objective of this study is to examine the efficacy of HD-tDCS to the preSMA/DACC region and its influence on verbal episodic memory in patients with MCI or dementia after 10 sessions of HD-tDCS. There will be three treatment arms: two active HD-tDCS (1 mA or 2 mA) and a sham group. A verbal episodic memory task will be completed at baseline, immediately following the last HD-tDCS session, and a 2-month follow-up.

DETAILED DESCRIPTION:
This is a pilot study being done to attempt to improve verbal episodic memory in persons with mild cognitive impairment (MCI) and dementia. Although the hippocampus is a brain structure most often associated with early deficits in MCI and dementia, the pre-supplemental motor area (preSMA) and dorsal anterior cingulate cortex (DACC) have been shown to play a role in verbal episodic memory for such patients. The purpose of this study is to examine the efficacy of high-definition transcranial direct current stimulation (HD-tDCS) to the preSMA/DACC region and its influence on verbal episodic memory in patients with MCI and dementia. Entraining the preSMA/DACC circuit with 10 sessions at one of two levels of HD-tDCS will allow the researchers to investigate whether neuromodulation may be used to improve verbal episodic memory. Participants will receive 10 sessions at one of two levels of active stimulation (1 mA or 2 mA anodal HD-tDCS targeting preSMA/DACC for 20 min) or sham across 2 weeks. The device is used to deliver high definition transcranial direct current stimulation to targeted regions. A verbal episodic memory task will be completed at baseline, immediately following the last HD-tDCS session, and a 2-month follow-up. The investigators plan to recruit English-speaking participants aged 50 years and older with MCI and dementia. Participants will be randomized into HD-tDCS conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 50 and older
2. Fluent in English
3. Active diagnosis of MCI or dementia

Exclusion Criteria:

1. Substance use disorder
2. Has metal fragments in head
3. Taking medications that may interact with the HD-tDCS effect (i.e., amphetamines, L-dopa, carbamazepine, sulpiride, pergolide, lorazepam, dextromethorphan, D-cycloserine, flunarizine, or ropinirole)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian LoBue, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LoBue C, Chiang HS, Salter A, McClintock S, Nguyen TP, Logan R, Smernoff E, Pandya S, Hart J. High definition transcranial direct current stimulation as an intervention for cognitive deficits in Alzheimer's dementia: A randomized controlled trial. J Prev Alzheimers Dis. 2025 Feb;12(2):100023. doi: 10.1016/j.tjpad.2024.100023. Epub 2025 Jan 1. PMID 39863318

RESULTS

PARTICIPANT FLOW:
Period: Assigned to Treatment
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Started | 6 | 13 | 14
Assigned to Treatment With Mild Cognitive Impairment | 1 | 3 | 0
Assigned to Treatment With Alzheimer Dementia | 5 | 10 | 14
Completed | 6 | 13 | 14
Not Completed | 0 | 0 | 0
Period: Started Treatment
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Started | 5 | 12 | 13
Started Treatment With Diagnosis of Mild Cognitive Impairment | 0 | 3 | 0
Started Treatment With Diagnosis of Alzheimer Dementia | 5 | 9 | 13
Completed | 5 | 12 | 9
Not Completed | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 1
Period: Follow-Up at 2 Months
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Started | 5 | 12 | 9
Completed | 4 | 12 | 9
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Analysis - Primary Outcomes Available
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Started | 5 | 12 | 9
Outcomes Available With Mild Cognitive Impairment | 0 | 2 | 0
Outcomes Available With Alzheimer Dementia | 5 | 10 | 9
Completed | 5 | 9 | 9
Not Completed | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Participants with mild cognitive impairment were not analyzed given the limited numbers that were recruited, allocated to treatment, and with data on outcome measures.
Groups:
- Sham Group: sham HD-tDCS for 20 minutes, meaning no stimulation.
- Active Stimulation at 1mA: 1 mA active HD-tDCS for 20 minutes.
- Active Stimulation at 2mA: 2 mA active HD-tDCS for 20 minutes.
- Total: Total of all reporting groups
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA | Total
Number analyzed (Participants) | 5 | 9 | 9 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (9.0) | 74.0 (9.5) | 68.4 (7.8) | 70.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 11
  Male | 3 | 5 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 8 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 5 | 9 | 7 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 9 | 9 | 23
Education [Mean (Standard Deviation); unit: years] | 16.0 (3.2) | 14.3 (1.7) | 14.4 (2.4) | 14.7 (2.3)
Time since diagnosis [Mean (Standard Deviation); unit: years] — Population: Data missing for 3 participants
  years
    number analyzed (Participants) | 5 | 7 | 8 | 20
    (all) | 2.3 (1.0) | 3.4 (3.3) | 1.1 (1.0) | 2.3 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on the Rey Auditory Verbal Learning Test (RAVLT)
Description: The RAVLT is a verbal episodic memory task where a list of 15 words is read aloud for 5 consecutive trials followed by a 20 minute delayed recall trial. The number of items recalled immediately after each trial are summed to create a total learning score, ranging from 0-75. Also, the number of items recalled for the delayed trial are recorded as a delayed recall score, ranging from 0-15. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better episodic memory performance. Changes from baseline for the total learning and delayed recall scores at the last HD-tDCS session and the 2-month follow-up will be measured as the primary outcomes.
Time Frame: Baseline, immediately following last treatment session, and 2-months post treatment
Population: One participant lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Number analyzed (Participants) | 5 | 9 | 9
T-score on a scale
  RAVLT total learning Baseline | 13.8 (10.4) | 17.8 (11.2) | 18.0 (10.3)
  RAVLT Total Learning Immediate post-treatment | 13.4 (11.7) | 21.0 (9.7) | 21.9 (12.8)
  RAVLT Total Learning 2 months: number analyzed (Participants) | 4 | 9 | 9
  RAVLT Total Learning 2 months | 16.3 (5.6) | 23.3 (13.8) | 17.2 (11.0)
  RAVLT Delayed Baseline | 20.6 (0.9) | 24.4 (6.1) | 22.3 (2.7)
  RAVLT Delayed Immediate Post-treatment | 21.2 (1.8) | 24.0 (6.2) | 22.3 (1.8)
  RAVLT Delayed 2 Months: number analyzed (Participants) | 4 | 9 | 9
  RAVLT Delayed 2 Months | 21.8 (1.5) | 25.7 (10.1) | 21.1 (1.3)
Statistical Analysis 1: Comparison: Sham Group vs Active Stimulation at 1mA; RAVLT Total Learning; Test type: Superiority; p = 0.25, ANCOVA; Cohen's d = 0.93
Statistical Analysis 2: Comparison: Sham Group vs Active Stimulation at 2mA; RAVLT Total Learning; Test type: Superiority; p = 0.18, ANCOVA; Cohen's d = 0.69
Statistical Analysis 3: Comparison: Sham Group vs Active Stimulation at 1mA; RAVLT Delayed; Test type: Superiority; p = 0.48, ANCOVA; Cohen's d = 0.74
Statistical Analysis 4: Comparison: Sham Group vs Active Stimulation at 2mA; RAVLT Delayed; Test type: Superiority; p = 0.64, ANCOVA; Cohen's d = 0.19

2. Secondary Outcome: Change in Score on the Brief Visuospatial Memory Test-Revised (BVMT-R)
Description: The BVMT-R is a visual episodic memory task where 6 simple designs are shown for 10 seconds in a 2 x 3 matrix for 3 learning trials followed by a 25-minute delayed recall trial. The number of items recalled immediately after each trial are summed to create a total learning score, ranging from 0-36. Also, the number of items recalled for the delayed trial are recorded as a delayed recall score, ranging from 0-12. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better visual episodic memory performance. Changes from baseline for the total learning and delayed recall scores at the last HD-tDCS session and the 2-month follow-up will be measured.
Time Frame: Baseline, immediately following last treatment session, and 2-months post treatment
Population: One participant lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Number analyzed (Participants) | 5 | 9 | 9
T-score on a scale
  BVMT Total Learning Baseline | 20.8 (1.1) | 24.2 (8.9) | 21.7 (3.1)
  BVMT Total Learning Immediate Post-treatment | 22.8 (2.6) | 24.2 (5.2) | 21.1 (2.0)
  BVMT Total Learning 2 Months: number analyzed (Participants) | 4 | 9 | 9
  BVMT Total Learning 2 Months | 20.0 (0.0) | 24.6 (9.9) | 20.7 (1.0)
  BVMT Delayed Baseline | 21.4 (3.1) | 26.9 (12.7) | 20.3 (1.0)
  BVMT Delayed Immediate Posttreatment | 20.6 (1.3) | 24.7 (10.1) | 22.8 (5.2)
  BVMT Delayed 2 Months: number analyzed (Participants) | 4 | 9 | 9
  BVMT Delayed 2 Months | 20.3 (0.5) | 25.4 (11.5) | 21.1 (2.4)
Statistical Analysis 1: Comparison: Sham Group vs Active Stimulation at 1mA; BVMT total learning; Test type: Superiority; p = 0.98, ANCOVA; Cohen's d = 0.03
Statistical Analysis 2: Comparison: Sham Group vs Active Stimulation at 2mA; BVMT total learning; Test type: Superiority; p = 0.22, ANCOVA; Cohen's d = 0.86
Statistical Analysis 3: Comparison: Sham Group vs Active Stimulation at 1mA; BVMT delayed; Test type: Superiority; p = 0.97, ANCOVA; Cohen's d = 0.04
Statistical Analysis 4: Comparison: Sham Group vs Active Stimulation at 2mA; BVMT delayed; Test type: Superiority; p = 0.23, ANCOVA; Cohen's d = 0.69

3. Secondary Outcome: Change in Score on the Boston Naming Test Short Form
Description: The Boston Naming Test Short Form is a 30 item version of the task (odd and even item versions of the full test) and a measure of language. The subject is shown pictures of objects and is required to correctly name them as quickly as possible. The outcome measure for this task is the total number of correct responses, ranging from 0-30. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance. Changes from baseline to the last HD-tDCS session and the 2-month follow-up will be measured.
Time Frame: Baseline, immediately following last treatment session, and 2-months post treatment
Population: One participant lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Number analyzed (Participants) | 5 | 9 | 9
T-score on a scale
  Baseline | 30.6 (16.2) | 31.6 (8.1) | 30.1 (9.0)
  Immediate Posttreatment | 30.4 (14.9) | 31.5 (9.0) | 31.9 (8.1)
  2 Months: number analyzed (Participants) | 4 | 9 | 9
  2 Months | 39.5 (27.7) | 32.1 (8.5) | 27.6 (8.4)
Statistical Analysis 1: Comparison: Sham Group vs Active Stimulation at 1mA; Test type: Superiority; p = 0.94, ANCOVA; Cohen's d = 0.04
Statistical Analysis 2: Comparison: Sham Group vs Active Stimulation at 2mA; Test type: Superiority; p = 0.47, ANCOVA; Cohen's d = 0.42

4. Secondary Outcome: Change in Score on the Delis Kaplan Executive Function System (DKEFS) Phonemic Fluency
Description: The DKEFS phonemic verbal fluency task is a measure of language. The subject is required to name as many words as possible that begin with specified letters within 1 minute. Three different letter trials are completed. The outcome measure for this task is the total number of correct responses across the trials, ranging from 0-90. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance. Changes from baseline to the last HD-tDCS session and the 2-month follow-up will be measured.
Time Frame: Baseline, immediately following last treatment session, and 2-months post treatment
Population: One participant lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Number analyzed (Participants) | 5 | 9 | 9
T-score on a scale
  Baseline | 39.0 (13.7) | 37.5 (8.7) | 32.7 (14.5)
  Immediate Posttreatment | 33.6 (14.9) | 40.4 (9.7) | 35.9 (14.2)
  2 Months: number analyzed (Participants) | 4 | 9 | 9
  2 Months | 35.3 (11.0) | 41.7 (9.9) | 32.1 (12.3)
Statistical Analysis 1: Comparison: Sham Group vs Active Stimulation at 1mA; Test type: Superiority; p = 0.06, ANCOVA; Cohen's d = 1.49
Statistical Analysis 2: Comparison: Sham Group vs Active Stimulation at 2mA; Test type: Superiority; p = 0.07, ANCOVA; Cohen's d = 1.08

5. Secondary Outcome: Change in Score on the Delis Kaplan Executive Function System (DKEFS) Semantic Fluency
Description: The DKEFS semantic verbal fluency task is a measure of language and involves 3 conditions. The subject is required to name as many animals and people names as possible within 1 minute. The outcome measure for this task is the total number of correct responses for both conditions combined, ranging from 0-90. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance. Changes from baseline to the last HD-tDCS session and the 2-month follow-up will be measured.
Time Frame: Baseline, immediately following last treatment session, and 2-months post treatment
Population: One participant lost to follow-up
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Number analyzed (Participants) | 5 | 9 | 9
T-score on a scale
  Baseline | 24.2 (10.6) | 28.1 (6.4) | 24.9 (6.0)
  Immediate Posttreatment | 25.0 (15.7) | 30.9 (8.7) | 22.8 (5.6)
  2 Months: number analyzed (Participants) | 4 | 9 | 9
  2 Months | 24.5 (9.0) | 30.2 (13.1) | 23.9 (4.6)
Statistical Analysis 1: Comparison: Sham Group vs Active Stimulation at 1mA; Test type: Superiority; p = 0.61, ANCOVA; Cohen's d = 0.19
Statistical Analysis 2: Comparison: Sham Group vs Active Stimulation at 2mA; Test type: Superiority; p = 0.38, ANCOVA; Cohen's d = 0.68

6. Secondary Outcome: Change in Score on the Trail Making Test
Description: The Trail Making Test is a measure of cognitive flexibility and executive functions. The task requires the subject to as quickly as possible complete two conditions, involving number sequencing and then number-letter switching. The outcome measure for this task is the time in seconds to complete the number-letter switching condition, ranging from 15-300. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance. Changes from baseline to the last HD-tDCS session and the 2-month follow-up will be measured.
Time Frame: Baseline, immediately following last treatment session, and 2-months post treatment
Population: Several participants were unable to complete the test in the administration time due to the level of cognitive impairment. Thus, the test was discontinued for many participants, prohibiting scores to be derived for several in data analysis. Scores are therefore missing for these, and the number that was able to complete the test varied across conditions and time points.
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Number analyzed (Participants) | 5 | 9 | 9
T-score on a scale
  Baseline: number analyzed (Participants) | 4 | 6 | 8
  Baseline | 22.3 (19.1) | 31.3 (17.4) | 22.8 (9.9)
  Immediate Posttreatment: number analyzed (Participants) | 3 | 8 | 7
  Immediate Posttreatment | 28.0 (27.4) | 24.4 (14.8) | 20.6 (13.2)
  2 Months: number analyzed (Participants) | 4 | 8 | 9
  2 Months | 24.5 (20.4) | 28.5 (15.8) | 19.7 (10.5)

7. Secondary Outcome: Change in Score on the Southwestern Assessment of Processing Speed
Description: The Southwestern Assessment of Processing Speed is a measure of psychomotor processing speed. The subject is required to transcribe numbers to their corresponding written symbol as quickly as possible within 60 seconds. The outcome measure for this task is the total number of correct responses, ranging from 0-75. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance. Changes from baseline to the last HD-tDCS session and the 2-month follow-up will be measured.
Time Frame: Baseline, immediately following last treatment session, and 2-months post treatment
Population: One participant lost to follow-up. Data missing for this measure on one participant in active 2 mA group.
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Number analyzed (Participants) | 5 | 9 | 9
T-score on a scale
  Baseline | 27.6 (7.7) | 34.0 (14.0) | 26.1 (5.5)
  Immediate Posttreatment | 30.2 (10.1) | 31.0 (10.0) | 27.9 (8.8)
  2 Months: number analyzed (Participants) | 4 | 9 | 8
  2 Months | 27.8 (6.8) | 30.8 (9.3) | 29.1 (10.6)
Statistical Analysis 1: Comparison: Sham Group vs Active Stimulation at 1mA; Test type: Superiority; p = 0.11, ANCOVA; Cohen's d = 0.96
Statistical Analysis 2: Comparison: Sham Group vs Active Stimulation at 2mA; Test type: Superiority; p = 0.68, ANCOVA; Eta2 effect sizes produced from the pairwise comparisons were transformed to Cohen's d for examination of effect sizes. A small/weak effect size was demonstrated (Cohen's d = 0.10), when adjusting for baseline performance

8. Secondary Outcome: Change in Score on the DKEFS Color-Word Interference Test
Description: The DKEFS Color-Word Interference test is a measure of information processing speed and complex attention. The task requires the subject to as quickly as possible complete four conditions, involving color naming, word reading, response inhibition, and then switching back-and-forth between two response patterns. The outcome measures for this task was the response inhibition trial and the switching trial, which are scored as the time in seconds to complete the conditions, ranging from 20-180. Scores were converted to standardized scores (T-scores) using normative data, ranging from 2-86. Higher scores reflect better performance. Changes from baseline to the last HD-tDCS session and the 2-month follow-up will be measured.
Time Frame: Baseline, immediately following last treatment session, and 2-months post treatment
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: T-score on a scale
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
Number analyzed (Participants) | 5 | 9 | 9
T-score on a scale
  Baseline: number analyzed (Participants) | 4 | 7 | 6
  Baseline | 35.5 (21.8) | 25.1 (10.6) | 35.0 (14.4)
  Immediate Posttreatment: number analyzed (Participants) | 3 | 7 | 6
  Immediate Posttreatment | 29.7 (20.2) | 30.3 (12.9) | 34.2 (13.8)
  2 Months: number analyzed (Participants) | 4 | 8 | 5
  2 Months | 25.0 (14.0) | 28.3 (14.3) | 36.4 (14.0)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the start of assigned treatments (1 mA, 2 mA, and sham) through study completion. This involved collection of information about adverse effects daily at the beginning and end of each treatment session and then again at the 2-month visit.
Arm/Group | Sham Group | Active Stimulation at 1mA | Active Stimulation at 2mA
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/12 | 1/13
Other Adverse Events (participants affected / at risk) | 0/5 | 0/12 | 0/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Group (N=5) | Active Stimulation at 1mA (N=12) | Active Stimulation at 2mA (N=13)
Hospitalization (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — Patient with pre-existing cardiac condition discovered to have cardiac decline during a medical visit. Hospitalized and treated. Participant recovered well. Not considered related to the treatment protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT05270408/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT05270408/SAP_001.pdf